CLINICAL TRIAL: NCT00287482
Title: A Pilot Study of the Herbal Remedy Essiac (ESIAK ®) Versus Placebo in Improving the Quality of Life in Women Completing Adjuvant Treatment for Breast or Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancers.
Brief Title: Essiac (ESIAK) Versus Placebo to Improve Quality of Life in Transition in Women With Breast or Ovarian Cancer.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WIH042005
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: Treatment side effects; Quality of Life; Transition; Survivorship
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — Essiac

INTERVENTIONS:
Drug: Essiac

SUMMARY:
This is a pilot feasibility study being performed in women completing front-line treatment for breast or ovarian cancer. It is being done to evaluate whether or not an herbal combination known as Essiac (ESIAK) can improve the overall quality of life in these women as they transition from active treatment to follow-up, also known as the quality of life in transition. This information will be used to design a larger randomized trial.

DETAILED DESCRIPTION:
Complementary and Alternative medical (CAM) practices are "healthcare practices outside the realm of conventional medicine, which are yet to be validated using scientific methods". It encompasses a wide variety of behavioral (meditation, and spiritual practices) and clinical (herbal, acupuncture, and massage) techniques. Patients with chronic diseases including cancer tend to be very interested in these treatments and research involving CAM and their ability to improve quality of life are needed.

Women transitioning from active treatment for breast or ovarian cancer to surveillance (QOL-T) can experience physical and psychological distress, related to both treatment (fatigue, alopecia, and menopausal symptoms), and the diagnosis itself. Intervention during the critical time of transition from active therapy to follow-up may help patients to adjust to life after cancer treatment.

Essiac has been documented to be a popular form of herbal treatment in patients with cancer. Given its lack of reported side effects, we are interested in pursuing a formal evaluation of a Essiac in capsule formulation (ESIAK) in women surviving breast or ovarian cancers to evaluate its role in improving the overall quality of life following chemotherapy that often accompanies the end of adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria

* histologically documented diagnosis of infiltrating carcinoma of the breast or epithelial ovarian cancer. Given the similar clinical course of patients with fallopian tube and primary peritoneal carcinoma these patients will also be included in the study.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients must be either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Women of child-bearing potential must have a negative pregnancy test. If patients become pregnant during the course of the study, they will not be allowed to continue on the study.
* age ≥ 18 year-old
* Karnofsky performance status > 70%
* Ability to understand and willingness to sign informed consent
* Ability to perform and comply with follow-up on study
* No history of drug or alcohol abuse
* No antecedent history of depression prior to diagnosis of malignancy
* Must be ≥ 4 weeks from completion of chemotherapy or radiation therapy.
* Adequate hematopoietic function defined as: ANC ≥ 1500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 8 g/dL.
* Adequate renal and hepatic function defined as: Bilirubin ≤ 1.5 times upper limit of normal (ULN); SGOT ≤ 2.5 times ULN; Alkaline phosphatase ≤ 2.5 times ULN; Creatinine ≤ 2 times ULN.
* For patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer (EOC/FT/PPC): patients must have completed front-line treatment within 3 months of study entry and in a complete remission; Patients treated with neoadjuvant platinum-based chemotherapy prior to definitive surgery will be eligible; If serum CA-125 was elevated at diagnosis, it must also have normalized by end of treatment.
* For patients with breast cancer: patients must have completed adjuvant treatment with chemotherapy and radiation therapy (if recommended) within three months of study entry and deemed in complete remission; Treatment must have included adjuvant chemotherapy and radiation if recommended; Patients receiving neoadjuvant therapy will be eligible following completion of all adjuvant chemotherapy if indicated. Patients receiving hormonal therapy following chemotherapy will be eligible to participate. However, patients placed on Tamoxifen or other hormonal agents in lieu of chemotherapy will not be eligible.

Exclusion Criteria

* history or active secondary cancer within the last 5 years, except for superficial basal cell skin cancers
* residual chemotherapy-induced CTCv3.0 Grade 2 or greater non-hematologic toxicity
* they are unable to give informed consent
* they are unable to adhere to protocol
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* concurrent uncontrolled illness
* ongoing or active infection

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-10; Study Completion 2007-07

PRIMARY OUTCOMES:
Quality of Life

SECONDARY OUTCOMES:
Toxicity
Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Don S Dizon, MD, Principal Investigator — Women & Infants' Hospital of Rhode Island
Locations (1):
- Women & Infants' Hospital, Providence, Rhode Island, United States